CLINICAL TRIAL: NCT05281510
Title: A Phase 2a Study to Evaluate the Safety and Tolerability of a Regimen of Dual Anti-HIV Envelope Antibodies, VRC07-523LS and CAP256V2LS, in a Sequential Regimen With a TLR7 Agonist, Vesatolimod, in Early Antiretroviral-Treated HIV-1 Clade C-Infected Women
Brief Title: Study of VRC07-523LS, CAP256V2LS, and Vesatolimod, in Early Antiretroviral-treated HIV-1 Clade C-infected Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-382-5445; DOH-27-082021-8379 (Other: South African National Clinical Trials Registry)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — vesatolimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VRC07523LS + CAP256V2LS + Vesatolimod (VES) (Experimental): In Period 1 (Days 0-28), participants will receive ART through Period. On Days 0 & 14, participants will be administered VES 6mg orally and on Day 28, participants will be administered VES either 6 or 8mg orally. VRC07-523LS & CAP256V2LS 20mg/kg will be administered intravenously on Day 7. In Period 2 (Days 29-133 or until ART restart), participants will discontinue ART at Day 35 and remain off ART until reaching ART restart criteria. Participants will receive VES 6 or 8mg orally every 2 weeks from Day 29 or until plasma HIV-1 RNA is >=5000 copies/mL. In Period 3, (Days 134-336 or until ART restart), participants will continue ATI and no study treatment will be administered. In Period 4, (Days 337-413) participants who have not met ART restart criteria by Day 337 may choose to restart ART (Period 4a) or may choose to continue ATI until end of study (Period 4B). Any participants who meet ART restart criteria before the end of the study will remain in follow-up on ART (Period 4A).
  Interventions: Drug: Vesatolimod; Biological: VRC07523LS; Biological: CAP256V2LS

INTERVENTIONS:
Drug: Vesatolimod — Administered orally
  Other Names: GS-9620
Biological: VRC07523LS — Administered intravenously
Biological: CAP256V2LS — Administered intravenously

SUMMARY:
The goals of this clinical study are to learn more about the study drugs, VRC07-523LS, CAP256V2LS, and vesatolimod (VES) and how safe it is in women that have HIV and are on antiretroviral therapy (ART).

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years
* Females recruited from the Females Rising through Education, Support, and Health (FRESH) acute human immunodeficiency virus (HIV) infection cohort.
* Plasma human immunodeficiency -1 (HIV-1) ribonucleic acid (RNA) levels < 50 copies/mL at the screening visit.
* On antiretroviral (ART) regimen for ≥ 12 consecutive months prior to the screening visit.
* Have all the following laboratory values at the screening visit:

  * Hemoglobin ≥ 10.0 g/dL
  * White blood cells ≥ 2500 cells/μL
  * Platelets ≥ 125,000/mL
  * Absolute neutrophil counts ≥ 1000 cells/μL
  * Cluster of differentiation (CD)4+ T cell count ≥ 500 cells/μL
  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and bilirubin ≤ 2 × upper limit of normal (ULN)
  * Creatinine clearance ≥ 60 mL/min
* Women of childbearing potential to have documentation of agreement to follow study contraceptive requirements.
* Documented plasma HIV-1 RNA < 50 copies/mL for 12 consecutive months prior to the screening visit.
* In the judgment of the investigator, be in good general health.
* Documented history of viral sensitivity to VRC07-523LS or CAP256V2LS at the screening visit.

Key Exclusion Criteria:

* Have poor venous access that limits phlebotomy.
* Positive serum pregnancy test.
* Nursing participants.
* Females with coinfection and/or immunosuppression as described below:

  * Autoimmune disease requiring ongoing immunosuppression
  * Evidence of chronic hepatitis B virus (HBV) infection
  * Evidence of current hepatitis C virus (HCV) infection
  * Documented history of pre-ART CD4+ T cell count nadir < 200 cells/μL
  * History of opportunistic illness indicative of Stage 3 HIV
  * Acute febrile illness within 4 weeks prior to the first dose
* Have current alcohol or substance abuse judged by the investigator to potentially interfere with individual's compliance or individual's safety.
* Have been treated with systemic steroids, immunosuppressant therapies, or chemotherapeutic agents within 3 months prior to screening or are expected to receive these agents during the study.
* Have previous or current receipt of humanized or human monoclonal antibody (mAbs), or polyclonal immunoglobulin.
* Have previous history of an antidrug antibodies response to a therapeutic agent.
* Have previous receipt of an HIV vaccine.
* Received any vaccine or immunomodulatory medication within 4 weeks prior to screening.
* Have a history of any of the following:

  * Significant serious skin disease
  * Significant drug sensitivity or drug allergy
  * Known hypersensitivity to the study drugs, metabolites, or formulation excipients
  * Previous or current history of bleeding disorder, platelet disorder including unexplained acute or chronic thrombocytopenia
  * Autoimmune diseases including type 1 diabetes mellitus
* Have current Class C acquired immunodeficiency syndrome (AIDS)-defining condition.
* Have any serious or active medical or psychiatric illness that would interfere with participants treatment, assessment, or compliance with the protocol.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- FRESH Clinical Research Site: Females Rising through Education, Support and Health, Umlazi, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dong K, Asari V, Govender V, et al. Evaluation of 2 bNAbs plus vesatolimod in early-treated South African women with HIV-1 during ATI [CROI abstract 105]. Top Antivir Med. 2025;33:14
- [Background] Omange RW, Zhang L, Reddy K, et al. Presence of protective human leukocyte antigen class I and II is associated with improved analytical treatment interruption outcomes in a trial of vesatolimod and broadly neutralizing antibodies in South African women with early-treated clade C HIV-1. Presented at the Keystone HIV Cure: Antiretroviral Therapy-Free Control of HIV Infection Symposium; April 7-10, 2025; Durban, South Africa. Poster 2014.
- [Background] Dong K, SenGupta D, Gama L, et al. First HIV cure interventional trial in Africa with collaboration between academia, government, and industry. Presented at the 13th International AIDS Society (IAS) Conference on HIV Science; July 13-17, 2025; Kigali, Rwanda. ePoster EP1003.
- [Background] Cai Y, Zhang L, Omange RW, et al. Vesatolimod pharmacodynamic responses in a trial of vesatolimod and broadly neutralizing antibodies in early-treated South African women with clade C HIV-1. Presented at the 13th International AIDS Society (IAS) Conference on HIV Science; July 13-17, 2025; Kigali, Rwanda. Poster WEPEB018.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-382-5445

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a study site in South Africa.
Pre-assignment Details: 26 participants were screened.
Groups:
- VRC07-523LS + CAP256V2LS + Vesatolimod (VES): In Period 1 (Days 0 to 28), participants received antiretroviral therapy (ART) through Period. On Days 0 and 14, participants were administered VES 6mg orally and on Day 28, participants were administered VES either 6mg or 8mg orally. VRC07-523LS 20mg/kg & CAP256V2LS 20mg/kg were administered intravenously on Day 7. In Period 2 (Days 29 to 133 or until ART restart), participants discontinued ART at Day 35 and remained off ART until reaching ART restart criteria. Participants received VES 8mg orally every 2 weeks from Day 29 or until plasma human immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) was >=5000 copies/mL. In Period 3, (Days 134 to 336 or until ART restart), participants continued analytical treatment interruption (ATI) and no study treatment was administered. In Period 4, (Days 337-413) participants who had not met ART restart criteria by Day 337 either choose to restart ART (Period 4a) or choose to continue ATI until end of study (Period 4B). Any participants who met ART restart criteria before the end of the study remained in follow-up on ART (Period 4A).
Period: Overall Study
Arm/Group | VRC07-523LS + CAP256V2LS + Vesatolimod (VES)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- VRC07-523LS + CAP256V2LS + Vesatolimod (VES): In Period 1 (Days 0 to 28), participants received ART through Period. On Days 0 and 14, participants were administered VES 6mg orally and on Day 28, participants were administered VES either 6mg or 8mg orally. VRC07-523LS 20mg/kg & CAP256V2LS 20mg/kg were administered intravenously on Day 7. In Period 2 (Days 29 to 133 or until ART restart), participants discontinued ART at Day 35 and remained off ART until reaching ART restart criteria. Participants received VES 8mg orally every 2 weeks from Day 29 or until plasma HIV-1 RNA was >=5000 copies/mL. In Period 3, (Days 134 to 336 or until ART restart), participants continued ATI and no study treatment was administered. In Period 4, (Days 337 to 413) participants who had not met ART restart criteria by Day 337 either choose to restart ART (Period 4a) or choose to continue ATI until end of study (Period 4B). Any participants who met ART restart criteria before the end of the study remained in follow-up on ART (Period 4A).
Arm/Group | VRC07-523LS + CAP256V2LS + Vesatolimod (VES)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a study drug that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a study drug, whether or not the AE is considered related to the study drug. TEAE was defined as any AE that began on or after the study drug start date and no later than last exposure date after permanent discontinuation of study drug, or led to premature study drug discontinuation.
Time Frame: Up to 61.1 weeks
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- VRC07-523LS + CAP256V2LS + VES: In Period 1 (Days 0 to 28), participants received ART through Period. On Days 0 and 14, participants were administered VES 6mg orally and on Day 28, participants were administered VES either 6mg or 8mg orally. VRC07-523LS 20mg/kg & CAP256V2LS 20mg/kg were administered intravenously on Day 7. In Period 2 (Days 29 to 133 or until ART restart), participants discontinued ART at Day 35 and remained off ART until reaching ART restart criteria. Participants received VES 8mg orally every 2 weeks from Day 29 or until plasma HIV-1 RNA was >=5000 copies/mL. In Period 3, (Days 134 to 336 or until ART restart), participants continued ATI and no study treatment was administered. In Period 4, (Days 337 to 413) participants who had not met ART restart criteria by Day 337 either choose to restart ART (Period 4a) or choose to continue ATI until end of study (Period 4B). Any participants who met ART restart criteria before the end of the study remained in follow-up on ART (Period 4A).
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
percentage of participants | 95

2. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Graded Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was defined as an increase of at least 1 toxicity grade from baseline at any time postbaseline up to and including the last exposure date after permanent discontinuation of study drug. For maximum postbaseline toxicity grade, the most severe graded abnormality from all tests was counted for each participant.
  The severity grades were defined by Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities, Antiviral Toxicity Grading Scale, Version 01 April 2015. The CTCAE v5 grading scale was used to grade AEs determined to be cytokine release syndrome and infusion-related reactions.
  The grading for both scales are as follows: Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-Threatening, Grade 5 = Death.
Time Frame: Up to 61.1 weeks
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | VRC07-523LS + CAP256V2LS + Vesatolimod (VES)
Number analyzed (Participants) | 20
percentage of participants
  Any Grade 1 or Higher | 95
  Grade 1 | 20
  Grade 2 | 40
  Grade 3 | 35
  Grade 4 | 0

3. Secondary Outcome: Time to Viral Rebound (Confirmed ≥ 50 Copies/mL and ≥ 200 Copies/mL) Following ATI
Description: Virologic rebound is defined as at any visit a rebound in HIV-1 RNA to ≥ 50 copies/mL or ≥ 200 copies/mL, which is subsequently confirmed at the following scheduled or unscheduled visit. Time to rebound (in weeks) = (date of rebound or censoring date - ATI start date + 1) / 7.
Time Frame: Up to 56 weeks
Population: The Full Analysis Set included all participants who were enrolled into the study and had received at least 1 dose of study drug.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
weeks
  Confirmed ≥ 50 copies/mL | 11.00 [7.00 to 19.07]
  Confirmed ≥ 200 copies/mL | 11.00 [7.00 to 19.14]

4. Secondary Outcome: Change in Plasma Viral Load Set-point Following ATI
Description: Change in plasma viral load set-point between pre-ART value and prior to ART reinitiation following ATI was summarized.
  The pre-ART set point value is the HIV-RNA load count prior to start of initial ARV treatment recorded in the clinical database.
Time Frame: Pre-ART (Screening) and prior to ART reinitiation following ATI (Up to 56 weeks)
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 11
log10 copies/mL | -1.42 [-1.85 to -0.77]
Statistical Analysis 1: Comparison: VRC07-523LS + CAP256V2LS + VES; The comparison was between plasma viral HIV-1 RNA data at set-point and at pre-ART within the same treatment group; Test type: Other; p = 0.0020, Wilcoxon signed rank test

5. Secondary Outcome: Change From Baseline of Viral Load at the End of ATI
Description: Baseline value was the last available value collected on or prior to first dose of study drug.
Time Frame: Up to 48 weeks
Population: Participants in Full Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
log10 copies/mL | 2.96 [1.58 to 4.07]

6. Secondary Outcome: Time to ART Resumption Following ATI
Description: Time to ART resumption (in weeks) = (date of restart ART after ATI period start or censoring date - ATI start date + 1) / 7.
Time Frame: Up to 56 weeks
Population: Participants in full analysis set were analyzed.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
weeks | 24.21 [12.64 to 47.14]

7. Secondary Outcome: Pharmacokinetic (PK) Parameter of VES: Cmax
Description: Cmax is defined as maximum observed concentration of drug.
Time Frame: Day 1: Predose (≤ 5 minutes prior to dosing), 1, 2, 4, 8, 12, 24, and 48 hours postdose
Population: The VES PK Analysis Set included all participants who were enrolled and had received at least 1 dose of VES and for whom PK concentrations of analyte VES were available.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
pg/mL | 6350 (4220)

8. Secondary Outcome: PK Parameter of VES: Tmax
Description: Tmax is defined as time (observed time point) of Cmax.
Time Frame: Day 1: Predose (≤ 5 minutes prior to dosing), 1, 2, 4, 8, 12, 24, and 48 hours postdose
Population: Participants in VES PK Analysis Set were analyzed.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
hours (h) | 2.00 [0.833 to 8.00]

9. Secondary Outcome: PK Parameter of VES: Clast
Description: Clast is defined as last observed quantifiable concentration of the drug.
Time Frame: Day 1: Predose (≤ 5 minutes prior to dosing), 1, 2, 4, 8, 12, 24, and 48 hours postdose
Population: Participants in VES PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
pg/mL | 279 (177)

10. Secondary Outcome: PK Parameter of VES: Tlast
Description: Tlast is defined as time (observed time point) of Clast.
Time Frame: Day 1: Predose (≤ 5 minutes prior to dosing), 1, 2, 4, 8, 12, 24, and 48 hours postdose
Population: Participants in VES PK Analysis Set were anlayzed.
Measure: Median (Full Range); unit: h
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
h | 48.0 [47.1 to 49.7]

11. Secondary Outcome: PK Parameter of VES: AUCinf
Description: AUCinf is defined as area under the concentration versus time curve extrapolated to infinite time, calculated as AUClast + (Clast/λz).
Time Frame: Day 1: Predose (≤ 5 minutes prior to dosing), 1, 2, 4, 8, 12, 24, and 48 hours postdose
Population: Participants in VES analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
h*pg/mL | 62700 (37700)

12. Secondary Outcome: PK Parameter of VES: AUClast
Description: AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration.
Time Frame: Day 1: Predose (≤ 5 minutes prior to dosing), 1, 2, 4, 8, 12, 24, and 48 hours postdose
Population: Participants in VES analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
h*pg/mL | 55500 (34200)

13. Secondary Outcome: PK Parameter of VES: AUCexp
Description: AUCexp is defined as AUC extrapolated between AUClast and AUCinf.
Time Frame: Day 1: Predose (≤ 5 minutes prior to dosing), 1, 2, 4, 8, 12, 24, and 48 hours postdose
Population: Participants in VES PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
percent | 12.4 (6.68)

14. Secondary Outcome: PK Parameter of VES: t1/2
Description: t1/2 is defined as estimate of the terminal elimination half-life of the drug, calculated by dividing the natural log of 2 by the terminal elimination rate constant (λz).
Time Frame: Day 1: Predose (≤ 5 minutes prior to dosing), 1, 2, 4, 8, 12, 24, and 48 hours postdose
Population: Participants in VES PK Analysis Set were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
h | 15.9 [10.4 to 27.0]

15. Secondary Outcome: PK Parameter of VES: CL/F
Description: CL/F is defined as apparent clearance following extravascular administration.
Time Frame: Day 1: Predose (≤ 5 minutes prior to dosing), 1, 2, 4, 8, 12, 24, and 48 hours postdose
Population: Participants in VES PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: Liters (L)/h
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
Liters (L)/h | 144 (112)

16. Secondary Outcome: PK Parameter of VES: Vz/F
Description: Vz/F is defined as apparent volume of distribution during the terminal phase following extravascular administration.
Time Frame: Day 1: Predose (≤ 5 minutes prior to dosing), 1, 2, 4, 8, 12, 24, and 48 hours postdose
Population: Participants with VES PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
L | 3810 (3650)

17. Secondary Outcome: PK Parameter of VRC07-523LS: Cmax
Description: Cmax is defined as maximum observed concentration of drug.
Time Frame: Day 7: Predose (0 hours), end of infusion, 1, 2, 4, and 8 hours after end of infusion, and then anytime on Days 8, 9, 14, 21, 28, 56, 84, 112, 133, 161, 189, 217, 245, 273, 301, 329, 343, 371, and 413
Population: The VRC07-523LS PK Analysis Set included all participants who were enrolled and had received at least 1 dose of VRC07-523LS and for whom PK concentrations of analyte VRC07-523LS were available. Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
µg/mL | 481 (83.5)

18. Secondary Outcome: PK Parameter of VRC07-523LS: Tmax
Description: Tmax is defined as time (observed time point) of Cmax.
Time Frame: as for outcome 17
Population: Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
h | 0.550 [0.467 to 4.83]

19. Secondary Outcome: PK Parameter of VRC07-523LS: Clast
Description: Clast is defined as last observed quantifiable concentration of the drug.
Time Frame: as for outcome 17
Population: Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
µg/mL | 3.51 (2.98)

20. Secondary Outcome: PK Parameter of VRC07-523LS: Tlast
Description: Tlast is defined as time (observed time point) of Clast.
Time Frame: as for outcome 17
Population: Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: day
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
day | 238 [147 to 336]

21. Secondary Outcome: PK Parameter of VRC07-523LS: AUCinf
Description: as for outcome 11
Time Frame: as for outcome 17
Population: Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
day*µg/mL | 7540 (1360)

22. Secondary Outcome: PK Parameter of VRC07-523LS: AUClast
Description: as for outcome 12
Time Frame: as for outcome 17
Population: Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
day*µg/mL | 7320 (1340)

23. Secondary Outcome: PK Parameter of VRC07-523LS: AUCexp
Description: AUCexp is defined as AUC extrapolated between AUClast and AUCinf.
Time Frame: as for outcome 17
Population: Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
percent | 2.94 (2.71)

24. Secondary Outcome: PK Parameter of VRC07-523LS: t1/2
Description: as for outcome 14
Time Frame: as for outcome 17
Population: Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: day
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
day | 41.9 [25.7 to 60.5]

25. Secondary Outcome: PK Parameter of VRC07-523LS: Clearance (CL)
Description: CL is defined as clearance following intravenous administration.
Time Frame: as for outcome 17
Population: Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
L/day | 0.198 (0.0513)

26. Secondary Outcome: PK Parameter of VRC07-523LS: Vss
Description: Vss is defined as the volume of distribution at steady-state following intravenous administration.
Time Frame: as for outcome 17
Population: Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: L
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
L | 11.5 (2.54)

27. Secondary Outcome: PK Parameter of VRC07-523LS: Vz
Description: Vz is defined as volume of distribution of the drug during the terminal phase after intravenous administration.
Time Frame: as for outcome 17
Population: Participants in VRC07-523LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
L | 12.0 (3.96)

28. Secondary Outcome: PK Parameter of CAP256V2LS: Cmax
Description: Cmax is defined as maximum observed concentration of drug.
Time Frame: as for outcome 17
Population: The CAP256V2LS PK Analysis Set included all participants who were enrolled and had received at least 1 dose of CAP256V2LS and for whom PK concentrations of analyte CAP256V2LS were available. Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
µg/mL | 644 (309)

29. Secondary Outcome: PK Parameter of CAP256V2LS: Tmax
Description: Tmax is defined as time (observed time point) of Cmax.
Time Frame: as for outcome 17
Population: Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
h | 1.50 [0.500 to 4.50]

30. Secondary Outcome: PK Parameter of CAP256V2LS: Clast
Description: Clast is defined as last observed quantifiable concentration of the drug.
Time Frame: as for outcome 17
Population: Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
µg/mL | 1.52 (0.493)

31. Secondary Outcome: PK Parameter of CAP256V2LS: Tlast
Description: Tlast is defined as time (observed time point) of Clast.
Time Frame: as for outcome 17
Population: Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: day
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
day | 172 [126 to 321]

32. Secondary Outcome: PK Parameter of CAP256V2LS: AUCinf
Description: as for outcome 11
Time Frame: as for outcome 17
Population: Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
day*µg/mL | 4290 (729)

33. Secondary Outcome: PK Parameter of CAP256V2LS: AUClast
Description: as for outcome 12
Time Frame: as for outcome 17
Population: Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
day*µg/mL | 4230 (710)

34. Secondary Outcome: PK Parameter of CAP256V2LS: AUCexp
Description: AUCexp is defined as AUC extrapolated between AUClast and AUCinf.
Time Frame: as for outcome 17
Population: Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
percent | 1.58 (0.452)

35. Secondary Outcome: PK Parameter of CAP256V2LS: t1/2
Description: as for outcome 14
Time Frame: as for outcome 17
Population: Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: day
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
day | 31.4 [20.2 to 77.8]

36. Secondary Outcome: PK Parameter of CAP256V2LS: CL
Description: CL is defined as clearance following intravenous administration.
Time Frame: as for outcome 17
Population: Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
L/day | 0.352 (0.116)

37. Secondary Outcome: PK Parameter of CAP256V2LS: Vz
Description: Vz is defined as volume of distribution of the drug during the terminal phase after intravenous administration.
Time Frame: as for outcome 17
Population: Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
L | 15.3 (3.72)

38. Secondary Outcome: PK Parameter of CAP256V2LS: Vss
Description: Vss is defined as the volume of distribution at steady-state after intravenous administration.
Time Frame: as for outcome 17
Population: Participants in CAP256V2LS PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 19
L | 10.6 (2.21)

39. Secondary Outcome: Percentage of Participants With Treatment-emergent Positive Anti-VRC07-523LS Antibodies
Time Frame: Prebaseline (Day -13) up to Day 413
Population: The VRC07-523LS Immunogenicity Analysis Set included all enrolled participants who received at least 1 dose of VRC07-523LS and have had at least 1 nonmissing value for the immunogenicity evaluation of interest (ie, anti-VRC07-523LS antibody).
Measure: Number; unit: percentage of participants
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
percentage of participants | 15.0

40. Secondary Outcome: Percentage of Participants With Treatment-emergent Positive Anti-CAP256V2LS Antibodies
Time Frame: Prebaseline (Day -13) up to Day 413
Population: The CAP256V2LS Immunogenicity Analysis Set included all enrolled participants who received at least 1 dose of CAP256V2LS and have had at least 1 nonmissing value for the immunogenicity evaluation of interest (ie, anti-CAP256V2LS antibody).
Measure: Number; unit: percentage of participants
Arm/Group | VRC07-523LS + CAP256V2LS + VES
Number analyzed (Participants) | 20
percentage of participants | 55

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events: Up to 61.1 weeks
Description: All-Cause Mortality: The Enrolled Analysis Set included all participants who were enrolled into the study.
  Adverse Events: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | VRC07-523LS + CAP256V2LS + VES
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VRC07-523LS + CAP256V2LS + VES (N=20)
Cellulitis (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Intentional self-injury (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VRC07-523LS + CAP256V2LS + VES (N=20)
Anaemia (Blood and lymphatic system disorders) | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 8
Eye irritation (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gingival swelling (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chest discomfort (General disorders) | 5
Chills (General disorders) | 3
Fatigue (General disorders) | 4
Influenza like illness (General disorders) | 3
Malaise (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 7
Swelling (General disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 2
Groin infection (Infections and infestations) | 1
Latent syphilis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 18
Haemoglobin decreased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 14
Paraesthesia (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Genital swelling (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT05281510/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT05281510/SAP_001.pdf